CLINICAL TRIAL: NCT01845675
Title: Temozolomide or Dacarbazine-based Chemotherapy Plus Endostatin in Advanced Pancreatic Neuroendocrine Tumor
Brief Title: Chemotherapy Plus Endostatin in Advanced Pancreatic Neuroendocrine Tumor
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Principal Investigator, YueJuan Cheng, attending medical oncologist, Peking Union Medical College Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TEPNET
Record Dates: First submitted 2013-04-29; First posted 2013-05-03 (Estimated); Last update posted 2017-04-13 (Actual); Status verified 2017-04

CONDITIONS: Advanced Well-differentiated Pancreatic Neuroendocrine Tumor
Keywords: temozolomide; endostatin; advanced; well-differentiated; pancreatic neuroendocrine tumor
MeSH Terms: conditions — Adenoma, Islet Cell | interventions — Temozolomide; Endostatins

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- temozolomide or dacarbazine-based chemotherapy, endostatin (Experimental): Endostatin 15mg/d，IV infusion, d1-d14 Temozolomide 150-200mg/m2/d，p.o., d1-d7 or dacarbazine 250mg/m2/d, IV infusion, d1-5, 5-FU 500mg/m2/d, IV infusion d1-5 Repeat every 3 weeks.
  Interventions: Drug: temozolomide or dacarbazine-based chemotherapy, endostatin

INTERVENTIONS:
Drug: temozolomide or dacarbazine-based chemotherapy, endostatin

SUMMARY:
Temozolomide or dacarbazine-based chemotherapy combined with endostatin have efficacy in well-differentiated pancreatic neuroendocrine tumor

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age and older
2. ECOG ≤2
3. Pathologically confirmed locally advanced or metastatic well-differentiated pancreatic neuroendocrine tumor.
4. Prior treatment with one-line chemotherapy is allowed, with the exception of prior treatment with temozolomide or dacarbazine or endostatin within the past 6 months
5. Disease progressed during or after last therapy
6. Minimum of 4 weeks since any major surgery, completion of radiation, or completion of all prior systemic anticancer therapy
7. Disease progressed within the past 12 months。
8. Patients must have at least one measurable site of disease according to RECIST1.1 criteria that has not been previously irradiated.
9. Adequate bone marrow, liver and renal function
10. Life expectancy 3 months or more
11. Patient informed consent。

Exclusion Criteria:

1. Concurrent use of Octreotide or other drug that may have efficacy in neuroendocrine tumor.
2. 2 or more lines of prior chemotherapy。
3. Patients who have any severe and/or uncontrolled medical conditions or other conditions that could affect their participation in the study
4. Uncontrolled infectious disease。
5. Other malignancies within the past 5 years except for adequately treated carcinoma of the cervix or basal or squamous cell carcinoma of the skin
6. Uncontrolled brain or leptomeningeal metastases
7. Patients with known hypersensitivity to temozolomide or endostatin。
8. Patient could not take tablets。

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2013-04; Primary Completion 2016-11-30 (Actual); Study Completion 2017-03-31 (Actual)

PRIMARY OUTCOMES:
overall response rate | up to 12 months

SECONDARY OUTCOMES:
progression free survival | From date of randomization until the date of first documented progression or date of death from any cause, whichever came first, assessed up to 24 months
toxicities | Number of participants with treatment-related adverse events as assessed by CTCAE v4.0

CONTACTS AND LOCATIONS:
Locations (1):
- Division of Medical Oncology, Peking Union Medical College Hospital, Beijing, China

IPD SHARING:
Plan to Share IPD: No